CLINICAL TRIAL: NCT02730000
Title: Cost-efficacy of Atraumatic Restorations (ART) Using Different Encapsulated Glass Ionomer Cement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Daniela Prócida Raggio, Associated Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RIVAART
Record Dates: First submitted 2016-02-22; First posted 2016-04-06 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Dental Caries
Keywords: Dental Atraumatic Restorative Treatment; Primary Teeth; Clinical Efficacy; Cost Analysis; Glass Ionomer Cement
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ART with Equia (Active Comparator): Occlusal-proximal restoration in primary molars using Equia (Easy/Quick/Unique/Intelligent/Aesthetic) from GC Corp, encapsulated, pre-dosed and mechanized handling.
  Interventions: Procedure: ART with Equia
- ART with Riva Self Cure (Experimental): Occlusal-proximal restoration in primary molars using Riva Self Cure from SDI, encapsulated, pre-dosed and mechanized handling.
  Interventions: Procedure: ART with Riva Self Cure

INTERVENTIONS:
Procedure: ART with Equia — Occlusal-proximal ART restorations in primary molars using Equia (Easy/Quick/Unique/ Intelligent/Aesthetic) will be performed. No local anesthesia will be used. Infected carious tissue will be removed with hand instruments, and the cavities restored with GIC (Glass Ionomer Cement). The cavity will be filled with GIC. After the press-finger technique, the excess of material will be removed and occlusion will be checked.
  Arms: ART with Equia
Procedure: ART with Riva Self Cure — Occlusal-proximal ART restorations in primary molars using Riva Self Cure will be performed. No local anesthesia will be used. Infected carious tissue will be removed with hand instruments, and the cavities restored with GIC (Glass Ionomer Cement). The cavity will be filled with GIC. After the press-finger technique, the excess of material will be removed and occlusion will be checked.
  Arms: ART with Riva Self Cure

SUMMARY:
Given the clinical damage caused by errors commonly made during the dosage and handling of glass ionomer cement (GIC) of high viscosity powder-liquid type, the use of encapsulated ionomer has been recommended for final restorations. However, the initial cost of the encapsulated MIC is higher when compared to the material handled manually. The objective of this randomized study is to (1) reveal cost-effective in the long run, the encapsulated CIV Riva Self Cure and Equia used as a restorative material in atraumatic restorations (Atraumatic Restorative Treatment), (2) assess whether the type of cavity (occlusal and occlusal-proximal) influences the longevity of atraumatic restorations using encapsulated IC, (3) assess whether the child's caries experience influences the longevity of atraumatic restorations with GIC encapsulated. Children, ages 3 and 7, will be selected in the Tietê-SP municipality. Randomization will be performed in a stratified manner by the conditions: type of cavity and caries experience. 122 ART restorations are performed using encapsulated CIV - Riva Self Cure - SDI and Equia -CG Corp. The restorations will be evaluated after 6, 12 and 18 months by two trained examiners blind to the groups (intra- and inter-rater agreement above 0.7). To verify the survival of the restorations will be used Kaplan-Meier survival analysis and log-rank test. To evaluate the association between longevity and variable Cox regression test will be applied. For the cost analysis will be used analysis of variance.

DETAILED DESCRIPTION:
Given the clinical damage caused by errors commonly made during the dosage and handling of glass ionomer cement (GIC) of high viscosity powder-liquid type, the use of encapsulated ionomer has been recommended for final restorations. However, the initial cost of the encapsulated MIC is higher when compared to the material handled manually. The objective of this randomized study is to (1) reveal cost-effective in the long run, the encapsulated CIV Riva Self Cure and Equia used as a restorative material in atraumatic restorations (Atraumatic Restorative Treatment), (2) assess whether the type of cavity (occlusal and occlusal-proximal) influences the longevity of atraumatic restorations using encapsulated IC, (3) assess whether the child's caries experience influences the longevity of atraumatic restorations with GIC encapsulated. Children, ages 3 and 7, will be selected in the Tietê-SP municipality. Randomization will be performed in a stratified manner by the conditions: type of cavity and caries experience. 122 ART restorations are performed using encapsulated CIV - Riva Self Cure - SDI and Equia -CG Corp. The restorations will be evaluated after 6, 12 and 18 months by two trained examiners blind to the groups (intra- and inter-rater agreement above 0.7).

ELIGIBILITY:
Inclusion Criteria:

* Children aging between 4 and 8 years
* presenting good health conditions
* whose parents or legal guardians accept and sign the consent form
* with at least one occlusal proximal caries lesion in primary molars
* only occlusal-proximal surfaces with caries lesions with dentin involvement

Exclusion Criteria:

* severe behavioral issues
* presence of fistula or abscess near the selected tooth
* presence of pulp exposure in the selected tooth
* presence of mobility in the selected tooth

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 148 (Actual)
Dates: Start 2016-07; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Longevity of atraumatic restoration | up to 24 months
  The treatments will be classified as successful when they present a clinical satisfactory aspect. Otherwise, "minor failure" will be analyzed. "Minor failures" are those in which there is a defect in the restoration/crown, but it does not interfere with the tooth health.

SECONDARY OUTCOMES:
Cost-efficacy assessment | an average of 24 months
  Treatment costs will be calculated considering professional costs and procedure costs. In order to calculate the professional cost the time spent in each session will be converted in hours and multiplied by the medium income of the dentist per hour as related by the Brazilian Ministry of Labour and Employment ($36,23). On the other hand, to estimate the procedure cost, it will be considered both variable cost, which includes electricity and equipment depreciation, and materials cost. To calculate the equipment depreciation (peripherals, dental chair and instrumental), the investigators will consider their price, the lifespan of five years and a monthly use of 160 hours, using an estimate value per hour of $1,81. All materials used in each procedure will have their specifications and quantity registered. Prices will be inferences from the market value converted in US Dollars and obtained by the medium of the values from different places that commercialized the referred products.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela P Raggio, Professor, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bonifacio CC, Hesse D, de Oliveira Rocha R, Bonecker M, Raggio DP, van Amerongen WE. Survival rate of approximal-ART restorations using a two-layer technique for glass ionomer insertion. Clin Oral Investig. 2013 Sep;17(7):1745-50. doi: 10.1007/s00784-012-0859-1. Epub 2012 Oct 11. PMID 23053709
- [Result] Bonifacio CC, Kleverlaan CJ, Raggio DP, Werner A, de Carvalho RC, van Amerongen WE. Physical-mechanical properties of glass ionomer cements indicated for atraumatic restorative treatment. Aust Dent J. 2009 Sep;54(3):233-7. doi: 10.1111/j.1834-7819.2009.01125.x. PMID 19709111
- [Result] da Franca C, Colares V, Van Amerongen E. Two-year evaluation of the atraumatic restorative treatment approach in primary molars class I and II restorations. Int J Paediatr Dent. 2011 Jul;21(4):249-53. doi: 10.1111/j.1365-263X.2011.01125.x. Epub 2011 Mar 15. PMID 21401749
- [Result] de Amorim RG, Leal SC, Frencken JE. Survival of atraumatic restorative treatment (ART) sealants and restorations: a meta-analysis. Clin Oral Investig. 2012 Apr;16(2):429-41. doi: 10.1007/s00784-011-0513-3. Epub 2011 Jan 28. PMID 21274581
- [Result] Deepa G, Shobha T. A clinical evaluation of two glass ionomer cements in primary molars using atraumatic restorative treatment technique in India: 1 year follow up. Int J Paediatr Dent. 2010 Nov;20(6):410-8. doi: 10.1111/j.1365-263X.2010.01067.x. PMID 20642467
- [Result] Dowling AH, Fleming GJ. Are encapsulated anterior glass-ionomer restoratives better than their hand-mixed equivalents? J Dent. 2009 Feb;37(2):133-40. doi: 10.1016/j.jdent.2008.10.006. Epub 2008 Dec 6. PMID 19059689
- [Result] Frencken JE, Van 't Hof MA, Van Amerongen WE, Holmgren CJ. Effectiveness of single-surface ART restorations in the permanent dentition: a meta-analysis. J Dent Res. 2004 Feb;83(2):120-3. doi: 10.1177/154405910408300207. PMID 14742648
- [Result] Gibson G, Jurasic MM, Wehler CJ, Jones JA. Supplemental fluoride use for moderate and high caries risk adults: a systematic review. J Public Health Dent. 2011 Summer;71(3):171-84. PMID 21972457
- [Result] Harris R, Gamboa A, Dailey Y, Ashcroft A. One-to-one dietary interventions undertaken in a dental setting to change dietary behaviour. Cochrane Database Syst Rev. 2012 Mar 14;2012(3):CD006540. doi: 10.1002/14651858.CD006540.pub2. PMID 22419315
- [Result] Holmgren CJ, Lo EC, Hu D, Wan H. ART restorations and sealants placed in Chinese school children--results after three years. Community Dent Oral Epidemiol. 2000 Aug;28(4):314-20. doi: 10.1034/j.1600-0528.2000.280410.x. PMID 10901411
- [Result] Kawai Y, Murakami H, Takanashi Y, Lund JP, Feine JS. Efficient resource use in simplified complete denture fabrication. J Prosthodont. 2010 Oct;19(7):512-6. doi: 10.1111/j.1532-849X.2010.00628.x. Epub 2010 Aug 16. PMID 20723019
- [Result] Kemoli AM, van Amerongen WE. Influence of the cavity-size on the survival rate of proximal ART restorations in primary molars. Int J Paediatr Dent. 2009 Nov;19(6):423-30. doi: 10.1111/j.1365-263X.2009.01013.x. Epub 2009 Sep 1. PMID 19732191
- [Result] Kemoli AM, Opinya GN, van Amerongen WE, Mwalili SM. Two-year survival rates of proximal atraumatic restorative treatment restorations in relation to glass ionomer cements and Postrestoration meals consumed. Pediatr Dent. 2011 May-Jun;33(3):246-51. PMID 21703078
- [Result] Mickenautsch S, Yengopal V, Banerjee A. Atraumatic restorative treatment versus amalgam restoration longevity: a systematic review. Clin Oral Investig. 2010 Jun;14(3):233-40. doi: 10.1007/s00784-009-0335-8. Epub 2009 Aug 18. PMID 19688227
- [Result] van Duinen RN, Kleverlaan CJ, de Gee AJ, Werner A, Feilzer AJ. Early and long-term wear of 'fast-set' conventional glass-ionomer cements. Dent Mater. 2005 Aug;21(8):716-20. doi: 10.1016/j.dental.2004.09.007. PMID 16026667
- [Result] Mitchell CA, Orr JF, Russell MD. Capsulated versus hand-mixed glass-ionomer luting cements for post retention. J Dent. 1998 Jan;26(1):47-51. doi: 10.1016/s0300-5712(96)00079-6. PMID 9479925
- [Result] Nyvad B, Machiulskiene V, Baelum V. Reliability of a new caries diagnostic system differentiating between active and inactive caries lesions. Caries Res. 1999 Jul-Aug;33(4):252-60. doi: 10.1159/000016526. PMID 10343087
- [Result] Raggio DP, Hesse D, Lenzi TL, Guglielmi CA, Braga MM. Is Atraumatic restorative treatment an option for restoring occlusoproximal caries lesions in primary teeth? A systematic review and meta-analysis. Int J Paediatr Dent. 2013 Nov;23(6):435-43. doi: 10.1111/ipd.12013. Epub 2012 Nov 28. PMID 23190278
- [Result] Roeleveld AC, van Amerongen WE, Mandari GJ. Influence of residual caries and cervical gaps on the survival rate of Class II glass ionomer restorations. Eur Arch Paediatr Dent. 2006 Jun;7(2):85-91. doi: 10.1007/BF03320820. PMID 17140533
- [Result] Smales RJ, Yip HK. The atraumatic restorative treatment (ART) approach for the management of dental caries. Quintessence Int. 2002 Jun;33(6):427-32. PMID 12073723
- [Result] Takanashi Y, Penrod JR, Lund JP, Feine JS. A cost comparison of mandibular two-implant overdenture and conventional denture treatment. Int J Prosthodont. 2004 Mar-Apr;17(2):181-6. PMID 15119869
- [Result] van 't Hof MA, Frencken JE, van Palenstein Helderman WH, Holmgren CJ. The atraumatic restorative treatment (ART) approach for managing dental caries: a meta-analysis. Int Dent J. 2006 Dec;56(6):345-51. doi: 10.1111/j.1875-595x.2006.tb00339.x. PMID 17243467
- [Result] Yu C, Gao XJ, Deng DM, Yip HK, Smales RJ. Survival of glass ionomer restorations placed in primary molars using atraumatic restorative treatment (ART) and conventional cavity preparations: 2-year results. Int Dent J. 2004 Feb;54(1):42-6. doi: 10.1111/j.1875-595x.2004.tb00251.x. PMID 15005472
- [Result] Walsh T, Worthington HV, Glenny AM, Appelbe P, Marinho VC, Shi X. Fluoride toothpastes of different concentrations for preventing dental caries in children and adolescents. Cochrane Database Syst Rev. 2010 Jan 20;(1):CD007868. doi: 10.1002/14651858.CD007868.pub2. PMID 20091655
- [Derived] Garbim JR, Saihara CS, Olegario IC, Hesse D, Araujo MP, Bonifacio CC, Braga MM, Raggio DP. 2-year survival and cost analysis of occlusoproximal ART restorations using encapsulated glass ionomer cement in primary molars: a randomized controlled trial. BMC Oral Health. 2024 Jun 1;24(1):647. doi: 10.1186/s12903-024-04357-9. PMID 38824540